CLINICAL TRIAL: NCT01025258
Title: Improving Adherence and Clinical Outcomes of Cystic Fibrosis Patients Through a Collaborative Active Intervention Program of a Multidisciplinary Team
Brief Title: Improving Adherence and Clinical Outcome in Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ori Efrati, Head of Pediatric Pulmonary Dept, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7380-OE-CTIL
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Medication Adherence; Multidisciplinary Team; Clinical Outcomes
MeSH Terms: conditions — Cystic Fibrosis; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- frequent clinic visits (Active Comparator)
  Interventions: Behavioral: Frequent Scheduled CF clinic visits; Behavioral: frequent telephone calls to patients pre and post visits to the clinic

INTERVENTIONS:
Behavioral: Frequent Scheduled CF clinic visits — Mandatory scheduled visit at the CF clinic every 1-2 months or sooner, if needed, for an evaluation by a a specialized CF team member such as: a pulmonary physician, a gastroenterologist, a dietitian, a clinical pharmacist
Behavioral: frequent telephone calls to patients pre and post visits to the clinic — Frequent telephone calls for monitoring, educating and identifying barriers in adherence will be made by a designated CF team member such as the CF nurse or the CF clinical pharmacist.

SUMMARY:
The purpose of this study is to assess the impact of a collaborative active intervention program of a multi-disciplinary team on improving adherence to chronic medications and improve clinical outcomes in CF patients.

DETAILED DESCRIPTION:
Cystic fibrosis is a life-threatening hereditary multi-system disease predominantly affecting the pancreas and lungs. Advances in treatment have led to significant improvements in prognosis though this depends crucially upon adherence to treatment.

It has been demonstrated in chronic conditions that improving medication adherence can improve clinical outcome, though it can be a difficult and complex task.

This is the first trial assessing the impact of a collaborative active intervention program of a multi disciplinary team in improving adherence to specific chronic medications and improving clinical outcomes in CF patients.

The trial will be divided into two parts:

First Part The first part of the trial will be a retrospective one in which data will be collected at baseline, from eligible patient files and patients' pharmacy records receiving standard care for the past 12 months.

Second Part The second part of the trial will be an active interventional prospective one and will be conducted for 12 months. The active intervention will be composed of series of visits of patients attending the clinic every 2 months (or sooner, if needed) in which a specialized CF team member will follow on the progress of the patient in his field of expertise. Furthermore, frequent telephone calls for monitoring, educating and identifying barriers in adherence will be made by a designated team member such as the CF nurse or the CF clinical pharmacist.

On identifying problems concerning medication adherence (such as: difficulties receiving medications from the sick fund, unwillingness to do inhaled medications because of allegedly side effects, difficulties in swallowing pills, etc.) solutions will be suggested by the CF team members and will be examined accordingly on the following visits.

Adherence to specific chronic medications will be determined by a short self reported questionnaire, a structured interview with the clinical pharmacist and prescriptions refill history obtained from pharmacy records in every visit to the clinical pharmacist.

Outcomes will be measured from patient's hospital records at baseline, 6 months and 12 months from the starting point. Measured clinical outcomes will be: PFTs, number of hospital admissions, number of exacerbations, number of IV courses, time between each exacerbation, inflammatory markers, BMI, HRQoL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of Cystic fibrosis at all ages.
2. CF patients that should be treated with one or more of these chronic medications: Tobi (Tobramycin), Coliracin (Colistin), Pulmozyme (Dornase Alpha), Hypertonic Saline (HS), Creon (pancreatic enzymes), AquaADEKs (Multivitamin).
3. Patients willing to participate in a trial.
4. Presence of a parent/guardian capable of providing informed consent.
5. Patients attending CF clinic at least once every 12 months.

Exclusion Criteria:

1. Absence of a parent/guardian or unwillingness to provide permission.
2. Potential participant declines to provide assent.
3. Transplant patients.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine whether a collaborative intervention program of a multi disciplinary team improves clinical outcomes such as: number of hospital admissions, number of IV ABx courses, and change in %FEV1, BMI. | 6 months, 12 months
To determine whether a collaborative intervention program of a multi disciplinary team improves adherence to routinely prescribed CF medications: Tobi, Pulmozyme, Colistine , HS, Creon and AquADEKs multivitamins. | 6 months, 12 months

SECONDARY OUTCOMES:
To determine whether a collaborative intervention program of a multi-disciplinary team improves health related quality of life. | 6 months, 12 months
To inspect whether improved adherence to medications during intensive care for 1 year in CF will reduce cytokines and inflammatory markers | 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ori Efrati, MD, Principal Investigator — Sheba Medical Center; Vardit M Kalamaro, BPharm, MSc, Study Director — The Israeli Cystic Fibrosis Foundation; Ran Nissan, Pharm D Student, Study Chair — Hebrew University of Jerusalem
Locations (1):
- Pediatric pulmonary unit, The Edmod and Lili Safra children's Hospital, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Kettler LJ, Sawyer SM, Winefield HR, Greville HW. Determinants of adherence in adults with cystic fibrosis. Thorax. 2002 May;57(5):459-64. doi: 10.1136/thorax.57.5.459. PMID 11978927
- [Background] Hofer M. Advanced chronic lung disease: need for an active interdisciplinary approach. Swiss Med Wkly. 2007 Nov 3;137(43-44):593-601. doi: 10.4414/smw.2007.11680. PMID 17990153